CLINICAL TRIAL: NCT00659932
Title: Dealing With Anxiety: A Pilot Cognitive Behavioural Program for Diabetic Clinic Outpatient Attendees
Brief Title: Dealing With Anxiety: A Cognitive Behavioural Program for Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hunter and New England Health (Other)
Responsible Party: Dr Kerry Bowen, Hunter and New England Health
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 02/03/13/3.18
Record Dates: First submitted 2008-04-14; First posted 2008-04-17 (Estimated); Last update posted 2008-04-17 (Estimated); Status verified 2007-12

CONDITIONS: Diabetes Mellitus Type 2
Keywords: diabetes; cognitive behavioural therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Immediate Cognitive behavioural therapy (CBT)
- 2 (Active Comparator)
  Interventions: Behavioral: Delayed CBT

INTERVENTIONS:
Behavioral: Immediate Cognitive behavioural therapy (CBT) — The Dealing with Anxiety CBT Group Program comprises 7 group sessions: an initial five hour session followed by 6 three hour sessions over a three month period
  Arms: 1
Behavioral: Delayed CBT — Commencement of the CBT Group Program is delayed 3 months
  Arms: 2

SUMMARY:
This study was designed to assess whether a cognitive behavior therapy (CBT) program for diabetes clinic patients was acceptable, improved quality of life and produced measurable change in levels of depression, anxiety and stress.

DETAILED DESCRIPTION:
Having co-morbid anxiety or depression makes it difficult to carry out the activities for diabetes selfcare. Psychological interventions have been shown to result in improvements in HbA1C and depression. Reports on psychosocial outcomes are conflicting and there are no studies of quality of life. Our diabetes outpatient population has a higher prevalence of anxiety and depression compared to the general public and this led to the development of a group CBT intervention designed to reduce anxiety as a co-morbidity of diabetes.

ELIGIBILITY:
Inclusion Criteria:

* Consenting attendees of the Hunter Area Diabetes Services RNH Diabetes Outpatient Clinic

Exclusion Criteria:

* Accessibility problems including:

  * limited English
  * developmental disability
  * physical immobility
  * geographical distance
  * extreme age/frailty

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2002-05; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

PRIMARY OUTCOMES:
Hemoglobin A1C (HbA1C) | 6 months

SECONDARY OUTCOMES:
Depression Anxiety Stress Scale (DASS) | 6 months
Diabetes Quality of Life (ADDQoL) | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Newcastle Hospital, Newcastle, New South Wales, Australia